CLINICAL TRIAL: NCT05414669
Title: The Effect of Allopurinol on Malondialdehyde, Nitric Oxide, Kidney Injury Molecule-1 Urine Levels, Resistive Index and Renal Elastography in Kidney Stone Patients After Extra Corporeal Shockwave Lithotripsy
Brief Title: Allopurinol Effect on MDA,NO,KIM-1 Urine Levels, RI and Renal Elastography in Kidney Stone Patients Post ESWL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanglah General Hospital (Other)
Responsible Party: Principal Investigator, Kadek Budi Santosa, Urologist, Sanglah General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020.03.1.0645
Record Dates: First submitted 2022-04-27; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi | interventions — Allopurinol; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Key envelope was kept by third party and will be opened once the data analysis is done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Allopurinol 300 mg was administered orally for a total of 3 days, starting from the day before ESWL
  Interventions: Drug: Allopurinol Tablet 300 mg
- Control Group (Placebo Comparator): Placebo was administered orally for a total of 3 days, starting from the day before ESWL
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Allopurinol Tablet 300 mg — Allopurinol 300mg was given orally for a total of 3 days, beginning a day before ESWL.
  Other Names: Allopurinol
  Arms: Interventional group
Drug: Control Group — Placebo was given orally for a total of 3 days, beginning a day before ESWL.
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
Extracorporeal shock wave lithotripsy (ESWL) is accepted as the first treatment choice for most urinary stones. Still, it has adverse effects on the kidneys. The mechanism underlying the shock wave induced renal injury is not entirely understood, and oxidative stress has been speculated to be involved in this process. The Investigator evaluated the role of allopurinol, which works as a xanthine oxidase inhibitor and free radical scavenger in renal protection against oxidative effects of ESWL. In a randomized, double-blind placebo-controlled trial, a total of 70 patients with renal stones undergoing ESWL were randomly assigned to 2 groups. Group 1 receive allopurinol, and group 2 receive a placebo. Allopurinol 300mg was given orally for a total of 3 days, beginning a day before ESWL. The urinary excretion of malondialdehyde (MDA), nitric oxide (NO), and kidney injury molecule-1 (KIM-1) were determined by quantitative double antibody sandwich direct ELISA at baseline before ESWL then repeatedly two h, and 24 h after ESWL. The resistive index (RI) change of the interlobar artery was asses along with the measurement of the shear wave velocity (SWV) in the focal zone of the treated kidney before, two weeks, and four weeks after ESWL. Multivariate analyses were performed using repeated measure ANOVA to control covariates.

DETAILED DESCRIPTION:
Subjects with kidney stones who met the criteria were given a detailed explanation about this study by the research team, then followed by signing the informed consent. History was taken along with physical examination, complete blood count, Bun, creatinine, uric acid, urinalysis and also anthropometric measurements (weight and height). Then each subjects got one of the intervention drugs, either allopurinol 300mg or placebo. Allopurinol 300 mg was finely grounded and put into gelatin capsules. The placebo was made by using Saccharum lactis material which was inserted into a gelatin capsule as well. The shape, color, texture, and weight of the placebo capsules were made the same as the drug allopurinol. Allopurinol capsules and placebo were made by the Pharmacy section of Sanglah Hospital.

Subjects were randomly allocated using a permuted block method into the allopurinol or placebo group. Each subject received one type of capsule consisting of 3 capsules containing 300 mg allopurinol or placebo taken the day before ESWL, 2 hours before ESWL, and the day after ESWL.

The study was conducted double-blind where the researcher, subject, data collector, outcome adjudicator, and data analyst did not know the type of treatment. Medicines are given in sealed envelopes using an undisclosed code that will be uncovered at the end of the study.

For the preparation of ESWL subjects; each subjects got infusion of 0.9% NaCl with 20 drops per minute, ondansetron 8 mg i.v., pethidine bolus 50 mg i.v., followed by drip pethidine 50 mg and ketorolac 30 mg given in 500 ml NaCl 0.9% with 20 drops of 20 drops per minute.

The Investigator performed ESWL using a Siemen litostar vario which uses an electromagnetic generator. The number of shock waves given is 2500-3000 shock waves per session. The given shock wave strength is slim to 2 J in the initial 200 shock wave followed by 3 to 3.5 J in the remainder of the shock wave. The given shock wave frequency is 60 x/minute.

Urine samples were taken aseptically using the mid-portion method in the amount of 10 ml for examination of biomarkers KIM-1, NO, and MDA one hour before ESWL. Furthermore, the urine sample was taken 10 ml two hours after ESWL and one day after ESWL. Examination time after ESWL is calculated from the end of the ESWL session.

RI examination and renal SWV elastography were performed one hour before ESWL, followed by two weeks and one month after ESWL by the same radiology specialist.

Subject compliance with medication is evaluated based on the number of capsules taken from the entire drug administered. If the number of capsules taken is less, the subject will be excluded from the analysis. Adverse events or drug side effects are defined as unexpected events during the study, such as experiencing procedure-related complications or being allergic to allopurinol. The Investigator evaluated the subjects every week after ESWL to assess tolerance and possible side effects.

If there was any drug side effects or serious adverse events(SAE), the subjects were reported to the ethics committee as soon as possible, less than 24 hours from the first time they were discovered, and actions were carried out as quickly as possible until the series of events ends. SAE was written in detail on the SAE form, including the following; when it was first discovered, the manifestation of the incident, the conditions before the incident, the handling of the event, and the outcome.

If the subject experiences side effects such as allergic reactions (redness of the skin, swelling of the eyes or mouth) and severe gastrointestinal disturbances (vomiting, diarrhea), the subject will be excluded from the analysis. The subject will also be excluded from the analysis if they experience complications related to ESWL procedure such as ureteral obstruction, pain (VAS > 5), or there were signs of infection. Subjects will be evaluated when visiting the hospital according to schedule, telephone contact, or by making a home visit.

The envelope of intervention data will be opened after data analysis, witnessed by an independent team, namely the Sanglah Hospital pharmacy and the Sanglah Hospital research division.

ELIGIBILITY:
Inclusion Criteria:

* Patient with renal stone who meet ESWL criteria
* Age 18 to 59 years old
* Consent to join this study

Exclusion Criteria:

* Patient with Diabetes Melitus
* Patient with hypertension
* Patient with Chronic Kidney Disease stage IV and stage V
* Patient with urinary tract infection
* Patient with obesity
* Patient with uric acid more than 9mg/dL

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Oxidative Stress | Two hours post-ESWL
  Level of Malondialdehyde (MDA), Nitric Oxide (NO), and Kidney Injury molecule-1 (KIM-1) in urine were determined by quantitative double antibody sandwich direct ELISA
Oxidative Stress | 24 hours post ESWL
  Level of Malondialdehyde (MDA), Nitric Oxide (NO), and Kidney Injury molecule-1 (KIM-1) in urine were determined by quantitative double antibody sandwich direct ELISA
Renal vascular and biophysical damage | Two weeks after ESWL
  Resistive Index (RI) change of the interlobar artery and elastography of the ipsilateral renal focal zone at ESWL
Renal vascular and biophysical damage | One month after ESWL
  Resistive Index (RI) change of the interlobar artery and elastography of the ipsilateral renal focal zone at ESWL

CONTACTS AND LOCATIONS:
Overall Officials: Kadek B Santosa, Urologist, Principal Investigator — Sanglah General Hospital
Locations (1):
- Sanglah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No
We are no going to share any individual participant data (IPD) considering Participant's Confidentiality.

REFERENCES:
- [Background] Acharya, C.R., Sharma, A.K., and Kantharia, N.D. 2015. Involvement of oxidative stress in patients of gout and antioxidant effect of allopurinol. International Journal of Medical Science and Public Health; 4(2): pp 168 -172
- [Background] Aksoy H, Aksoy Y, Turhan H, Keles S, Ziypak T, Ozbey I. The effect of shock wave lithotripsy on nitric oxide and malondialdehyde levels in plasma and urine samples. Cell Biochem Funct. 2007 Sep-Oct;25(5):533-6. doi: 10.1002/cbf.1349. PMID 16850521
- [Background] Denic A, Mathew J, Lerman LO, Lieske JC, Larson JJ, Alexander MP, Poggio E, Glassock RJ, Rule AD. Single-Nephron Glomerular Filtration Rate in Healthy Adults. N Engl J Med. 2017 Jun 15;376(24):2349-2357. doi: 10.1056/NEJMoa1614329. PMID 28614683
- [Background] Alirezaei, A., Argani, H., Asgharpour, M., Bahadorimonfared, A., and Bakhtiyari, M. 2017. An update on allopurinol and kidney failure; new trend for an old drug. J Renal Inj Prev; 6(4): pp 297-302
- [Background] Alessio HM. 2000. In: Handbook of oxidants and antioxidants in exercise. Hanninen O, Packy L, Sen CK, editors. Elsevier; Amsterdam; pp 115-128
- [Background] Asnita Arif, Nurlaily Idris, Bachtiar Murtala, Andi Alfian Z, Sri Asriyani, and Hasyim Kasim. 2019. The Correlation Between Renal Shear Wave Elastography with Estimated Glomerular FiltrationRate in Chronic Kidney Disease. Jurnal Kedokteran Brawijaya; 30(4): pp 287-292
- [Background] Berry CE, Hare JM. Xanthine oxidoreductase and cardiovascular disease: molecular mechanisms and pathophysiological implications. J Physiol. 2004 Mar 16;555(Pt 3):589-606. doi: 10.1113/jphysiol.2003.055913. Epub 2003 Dec 23. PMID 14694147
- [Background] Bonventre JV. Kidney injury molecule-1 (KIM-1): a urinary biomarker and much more. Nephrol Dial Transplant. 2009 Nov;24(11):3265-8. doi: 10.1093/ndt/gfp010. Epub 2009 Mar 23. No abstract available. PMID 19318357
- [Background] Bonventre JV. Primary proximal tubule injury leads to epithelial cell cycle arrest, fibrosis, vascular rarefaction, and glomerulosclerosis. Kidney Int Suppl (2011). 2014 Nov;4(1):39-44. doi: 10.1038/kisup.2014.8. PMID 26310195
- [Background] Brian R, Matlaga, Amy E. Krambeck, and James E. Lingeman. 2016. Surgical management of Upper Urinary Tract Calculi. Campbell-Walsh urology. Philadelphia: Elsevier; pp 1260-1276
- [Background] Burne-Taney MJ, Ascon DB, Daniels F, Racusen L, Baldwin W, Rabb H. B cell deficiency confers protection from renal ischemia reperfusion injury. J Immunol. 2003 Sep 15;171(6):3210-5. doi: 10.4049/jimmunol.171.6.3210. PMID 12960350
- [Background] Busti A.J. 2015. The Differences in the Mechanisms of Action Between Allopurineol and Febuxostat. Available at: http://www.ebmconsult.com/articles/allopurinol\ and febuxostat-zyloprim-uloric-uric-acid-gout-mechanism. Accesed 9th August 2016
- [Background] Chawla LS, Eggers PW, Star RA, Kimmel PL. Acute kidney injury and chronic kidney disease as interconnected syndromes. N Engl J Med. 2014 Jul 3;371(1):58-66. doi: 10.1056/NEJMra1214243. No abstract available. PMID 24988558
- [Background] Coca SG, Yusuf B, Shlipak MG, Garg AX, Parikh CR. Long-term risk of mortality and other adverse outcomes after acute kidney injury: a systematic review and meta-analysis. Am J Kidney Dis. 2009 Jun;53(6):961-73. doi: 10.1053/j.ajkd.2008.11.034. Epub 2009 Apr 5. PMID 19346042
- [Background] Dahlan, M. Sopiyudin. 2009. Besar Sampel dan Pengambilan Sampel, dalam Penelitian Kedokteran dan Kesehatan. Jakarta: Salemba Medika
- [Background] Clark DL, Connors BA, Evan AP, Willis LR, Handa RK, Gao S. Localization of renal oxidative stress and inflammatory response after lithotripsy. BJU Int. 2009 Jun;103(11):1562-8. doi: 10.1111/j.1464-410X.2008.08260.x. Epub 2009 Jan 20. PMID 19154498
- [Background] Day RO, Graham GG, Hicks M, McLachlan AJ, Stocker SL, Williams KM. Clinical pharmacokinetics and pharmacodynamics of allopurinol and oxypurinol. Clin Pharmacokinet. 2007;46(8):623-44. doi: 10.2165/00003088-200746080-00001. PMID 17655371
- [Background] de Geus HR, Betjes MG, Bakker J. Biomarkers for the prediction of acute kidney injury: a narrative review on current status and future challenges. Clin Kidney J. 2012 Apr;5(2):102-108. doi: 10.1093/ckj/sfs008. PMID 22833807
- [Background] Denise grotto, lucas santa maria, Juliana Valentini, clóvis paniz, and gabriela schmitt e solange cristina garcia. 2009. Importance of the Lipid peroxidation biomarkers and methodological aspects for malondialdehyde quantification. Quim. Nova; 32(1): pp 169-174
- [Background] De Rosa S, Antonelli M, Ronco C. Hypothermia and kidney: a focus on ischaemia-reperfusion injury. Nephrol Dial Transplant. 2017 Feb 1;32(2):241-247. doi: 10.1093/ndt/gfw038. PMID 28186567
- [Background] Devarajan P. Update on mechanisms of ischemic acute kidney injury. J Am Soc Nephrol. 2006 Jun;17(6):1503-20. doi: 10.1681/ASN.2006010017. Epub 2006 May 17. No abstract available. PMID 16707563
- [Background] Dinh QN, Drummond GR, Sobey CG, Chrissobolis S. Roles of inflammation, oxidative stress, and vascular dysfunction in hypertension. Biomed Res Int. 2014;2014:406960. doi: 10.1155/2014/406960. Epub 2014 Jul 20. PMID 25136585
- [Background] Eddy AA. Molecular basis of renal fibrosis. Pediatr Nephrol. 2000 Dec;15(3-4):290-301. doi: 10.1007/s004670000461. PMID 11149129
- [Background] Erol T, Tekin A, Katircibasi MT, Sezgin N, Bilgi M, Tekin G, Zumrutdal A, Sezgin AT, Muderrisoglu H. Efficacy of allopurinol pretreatment for prevention of contrast-induced nephropathy: a randomized controlled trial. Int J Cardiol. 2013 Aug 20;167(4):1396-9. doi: 10.1016/j.ijcard.2012.04.068. Epub 2012 May 8. PMID 22572633
- [Background] Fahmy N, Sener A, Sabbisetti V, Nott L, Lang RM, Welk BK, Mendez-Probst CE, MacPhee RA, VanEerdewijk S, Cadieux PA, Bonventre JV, Razvi H. Urinary expression of novel tissue markers of kidney injury after ureteroscopy, shockwave lithotripsy, and in normal healthy controls. J Endourol. 2013 Dec;27(12):1455-62. doi: 10.1089/end.2013.0188. Epub 2013 Nov 1. PMID 24180435
- [Background] Fegan JE, Husmann DA, Alexander ME, Feagins B, and Preminger GM. 2009. Preservation of renal architecture durineg extracorporeal shock wave lithotripsy. J Endourol/Endourol Soc; 5: pp 273-6
- [Background] Garg AX, Parikh CR. Yin and Yang: acute kidney injury and chronic kidney disease. J Am Soc Nephrol. 2009 Jan;20(1):8-10. doi: 10.1681/ASN.2008111197. Epub 2008 Dec 31. No abstract available. PMID 19118145
- [Background] George J, Struthers AD. Role of urate, xanthine oxidase and the effects of allopurinol in vascular oxidative stress. Vasc Health Risk Manag. 2009;5(1):265-72. doi: 10.2147/vhrm.s4265. Epub 2009 Apr 8. PMID 19436671
- [Background] Graham S, Day RO, Wong H, McLachlan AJ, Bergendal L, Miners JO, Birkett DJ. Pharmacodynamics of oxypurinol after administration of allopurinol to healthy subjects. Br J Clin Pharmacol. 1996 Apr;41(4):299-304. doi: 10.1046/j.1365-2125.1996.03116.x. PMID 8730975
- [Background] Girardi G, Berman J, Redecha P, Spruce L, Thurman JM, Kraus D, Hollmann TJ, Casali P, Caroll MC, Wetsel RA, Lambris JD, Holers VM, Salmon JE. Complement C5a receptors and neutrophils mediate fetal injury in the antiphospholipid syndrome. J Clin Invest. 2003 Dec;112(11):1644-54. doi: 10.1172/JCI18817. PMID 14660741
- [Background] Han WK, Bailly V, Abichandani R, Thadhani R, Bonventre JV. Kidney Injury Molecule-1 (KIM-1): a novel biomarker for human renal proximal tubule injury. Kidney Int. 2002 Jul;62(1):237-44. doi: 10.1046/j.1523-1755.2002.00433.x. PMID 12081583
- [Background] Hatipoglu NK, Evliyaoglu O, Isik B, Bodakci MN, Bozkurt Y, Sancaktutar AA, Soylemez H, Atar M, Penbegul N, Yunce M, Daggulli M. Antioxidant signal and kidney injury molecule-1 levels in shockwave lithotripsy induced kidney injury. J Endourol. 2014 Feb;28(2):224-8. doi: 10.1089/end.2013.0535. Epub 2013 Nov 9. PMID 24044353
- [Background] Hirschberg R. Wound healing in the kidney: complex interactions in renal interstitial fibrogenesis. J Am Soc Nephrol. 2005 Jan;16(1):9-11. doi: 10.1681/ASN.2004110901. Epub 2004 Dec 1. No abstract available. PMID 15574504
- [Background] Hobarth K, Maier A, Hofbauer J, Marberger M. Color flow Doppler sonography for extracorporeal shock wave lithotripsy. J Urol. 1993 Dec;150(6):1768-70. doi: 10.1016/s0022-5347(17)35890-1. PMID 8230499
- [Background] Kalluri R, Neilson EG. Epithelial-mesenchymal transition and its implications for fibrosis. J Clin Invest. 2003 Dec;112(12):1776-84. doi: 10.1172/JCI20530. PMID 14679171
- [Background] Kira VM, Fagundes DJ, Bandeira CO, Kaufman O, Fagundes AT, Ortiz V. Effects of repeated extracorporeal shock wave on kidney apoptosis of normal and diabetic rat. Int Braz J Urol. 2008 Jan-Feb;34(1):91-6. doi: 10.1590/s1677-55382008000100013. PMID 18341726
- [Background] Kostic D.a., Dimitrijevic D.S., Stojanovic G.S., Palic I.R., Dordevic A.S., and Ickovski J.D. 2015. Xanthine Oxidase: Isolation, Assays of Activity, and Inhibition. Journal of Chemistry; available at https://doi.org/10.1155/2015/294858
- [Background] Kou B, Ni J, Vatish M, Singer DR. Xanthine oxidase interaction with vascular endothelial growth factor in human endothelial cell angiogenesis. Microcirculation. 2008 Apr;15(3):251-67. doi: 10.1080/10739680701651495. PMID 18386220
- [Background] Kurt S, Tokgoz O, Tokgoz H, Voyvoda N. Evaluation of effects of Extracorporeal Shock Wave Lithotripsy on renal vasculature with Doppler ultrasonography. Med Ultrason. 2013 Dec;15(4):273-7. doi: 10.11152/mu.2013.2066.154.sk2. PMID 24286090
- [Background] Levey AS, Eckardt KU, Tsukamoto Y, Levin A, Coresh J, Rossert J, De Zeeuw D, Hostetter TH, Lameire N, Eknoyan G. Definition and classification of chronic kidney disease: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x. PMID 15882252
- [Background] Li B, Zhou W, Li P. Protective effects of nifedipine and allopurinol on high energy shock wave induced acute changes of renal function. J Urol. 1995 Mar;153(3 Pt 1):596-8. PMID 7861490
- [Background] Liu Y. Epithelial to mesenchymal transition in renal fibrogenesis: pathologic significance, molecular mechanism, and therapeutic intervention. J Am Soc Nephrol. 2004 Jan;15(1):1-12. doi: 10.1097/01.asn.0000106015.29070.e7. PMID 14694152
- [Background] Macias-Nunez JF, Revert M, Fiksen-Olsen M, Knox FG, Romero JC. Effect of allopurinol on the renovascular responses to adenosine. J Lab Clin Med. 1986 Jul;108(1):30-6. PMID 3519811
- [Background] Margaret S. Pearle, and Yair Lotan. 2016. Urineary Lithiasis; Etiology, Epidemiology, and Pathogenesis. Campbell-Walsh urology. Philadelphia: Elsevier, pp.1363-1391
- [Background] McClintock DS, Santore MT, Lee VY, Brunelle J, Budinger GR, Zong WX, Thompson CB, Hay N, Chandel NS. Bcl-2 family members and functional electron transport chain regulate oxygen deprivation-induced cell death. Mol Cell Biol. 2002 Jan;22(1):94-104. doi: 10.1128/MCB.22.1.94-104.2002. PMID 11739725
- [Background] McDonagh EM, Thorn CF, Callaghan JT, Altman RB, Klein TE. PharmGKB summary: uric acid-lowering drugs pathway, pharmacodynamics. Pharmacogenet Genomics. 2014 Sep;24(9):464-76. doi: 10.1097/FPC.0000000000000058. No abstract available. PMID 24915143
- [Background] Miller NL, Evan AP, Lingeman JE. Pathogenesis of renal calculi. Urol Clin North Am. 2007 Aug;34(3):295-313. doi: 10.1016/j.ucl.2007.05.007. PMID 17678981
- [Background] Munver R, Delvecchio FC, Kuo RL, Brown SA, Zhong P, Preminger GM. In vivo assessment of free radical activity during shock wave lithotripsy using a microdialysis system: the renoprotective action of allopurinol. J Urol. 2002 Jan;167(1):327-34. PMID 11743351
- [Background] Nakao T, Ushigome H, Nakamura T, Harada S, Koshino K, Suzuki T, Ito T, Nobori S, Yoshimura N. Evaluation of renal allograft fibrosis by transient elastography (Fibro Scan). Transplant Proc. 2015 Apr;47(3):640-3. doi: 10.1016/j.transproceed.2014.12.034. PMID 25891702
- [Background] Mercimek MN, Ender O. Effect of urinary stone disease and its treatment on renal function. World J Nephrol. 2015 May 6;4(2):271-6. doi: 10.5527/wjn.v4.i2.271. PMID 25949941
- [Background] Weimert NA, Tanke WF, Sims JJ. Allopurinol as a cardioprotectant during coronary artery bypass graft surgery. Ann Pharmacother. 2003 Nov;37(11):1708-11. doi: 10.1345/aph.1D023. PMID 14565806
- [Background] Kwon O, Hong SM, Ramesh G. Diminished NO generation by injured endothelium and loss of macula densa nNOS may contribute to sustained acute kidney injury after ischemia-reperfusion. Am J Physiol Renal Physiol. 2009 Jan;296(1):F25-33. doi: 10.1152/ajprenal.90531.2008. Epub 2008 Oct 29. PMID 18971208
- [Background] Ozkan F, Goya C, Yildiz S, Duymus M, Menzilcioglu SM, and Avcu S. 2016. Ultrasound elastography in kidney disease. In: Patel VB, Preedy VR (ed), Biomarkers in Kidney Disease, Biomarkers in Disease: Methods, Discoveries and Applications; pp 1052-1072
- [Background] Ozturk A, Grajo JR, Dhyani M, Anthony BW, Samir AE. Principles of ultrasound elastography. Abdom Radiol (NY). 2018 Apr;43(4):773-785. doi: 10.1007/s00261-018-1475-6. PMID 29487968
- [Background] Platt JF. Duplex Doppler evaluation of native kidney dysfunction: obstructive and nonobstructive disease. AJR Am J Roentgenol. 1992 May;158(5):1035-42. doi: 10.2214/ajr.158.5.1566663.
- [Background] Pocock J. Stuart. 2013. Clinical Trials a Practical Approach. New York: Jon Wiley and Son-Brisbane-Toronto
- [Background] Pozniak, M., and Allan, P. 2014. Clinical doppler ultrasound (3rd ed). Philadelphia: Chucill-Livingstone Elsevier; pp 193-213
- [Background] Pries AR, Kuebler WM. Normal endothelium. Handb Exp Pharmacol. 2006;(176 Pt 1):1-40. doi: 10.1007/3-540-32967-6_1. PMID 16999215
- [Background] Puddu P, Puddu GM, Cravero E, Vizioli L, Muscari A. Relationships among hyperuricemia, endothelial dysfunction and cardiovascular disease: molecular mechanisms and clinical implications. J Cardiol. 2012 May;59(3):235-42. doi: 10.1016/j.jjcc.2012.01.013. Epub 2012 Mar 6. PMID 22398104
- [Background] Rosenblum ER, Gavaler JS, Van Thiel DH. Lipid peroxidation: a mechanism for alcohol-induced testicular injury. Free Radic Biol Med. 1989;7(5):569-77. doi: 10.1016/0891-5849(89)90034-8. PMID 2693225
- [Background] Sagor MA, Tabassum N, Potol MA, Alam MA. Xanthine Oxidase Inhibitor, Allopurinol, Prevented Oxidative Stress, Fibrosis, and Myocardial Damage in Isoproterenol Induced Aged Rats. Oxid Med Cell Longev. 2015;2015:478039. doi: 10.1155/2015/478039. Epub 2015 Jun 7. PMID 26137187
- [Background] Santoso dan Singgih. 2016. Statistik Parametrik Konsep dan Aplikasi dengan SPSS. Edisi Revisi.Jakarta: Media Komputindo (Gramedia).
- [Background] Shao X, Tian L, Xu W, Zhang Z, Wang C, Qi C, Ni Z, Mou S. Diagnostic value of urinary kidney injury molecule 1 for acute kidney injury: a meta-analysis. PLoS One. 2014 Jan 3;9(1):e84131. doi: 10.1371/journal.pone.0084131. eCollection 2014. PMID 24404151
- [Background] Shaw CA, Taylor EL, Megson IL, Rossi AG. Nitric oxide and the resolution of inflammation: implications for atherosclerosis. Mem Inst Oswaldo Cruz. 2005 Mar;100 Suppl 1:67-71. doi: 10.1590/s0074-02762005000900012. Epub 2005 Jun 14. PMID 15962101
- [Background] Singh H, Panta OB, Khanal U, Ghimire RK. Renal Cortical Elastography: Normal Values and Variations. J Med Ultrasound. 2017 Oct-Dec;25(4):215-220. doi: 10.1016/j.jmu.2017.04.003. Epub 2017 May 31. PMID 30065495
- [Background] Singh, I. and Strandhoy, J W. 2012. Pathophysiology of Urineary Tract Obstruction. In: Wein, A.J. Kavoussi, L.R. Novick, A.C. Partin, A.W.Peters, C.A. Editors. Campbell-Walsh Urology, 10th Ed. Saunders. Esevier. Philadelphia
- [Background] Stamp LK, Day RO, Yun J. Allopurinol hypersensitivity: investigating the cause and minimizing the risk. Nat Rev Rheumatol. 2016 Apr;12(4):235-42. doi: 10.1038/nrrheum.2015.132. Epub 2015 Sep 29. PMID 26416594
- [Background] Thurston MM, Phillips BB, Bourg CA. Safety and efficacy of allopurinol in chronic kidney disease. Ann Pharmacother. 2013 Nov;47(11):1507-16. doi: 10.1177/1060028013504740. Epub 2013 Oct 9. PMID 24259601
- [Background] Toprak O, Cirit M, Esi E, Postaci N, Yesil M, Bayata S. Hyperuricemia as a risk factor for contrast-induced nephropathy in patients with chronic kidney disease. Catheter Cardiovasc Interv. 2006 Feb;67(2):227-35. doi: 10.1002/ccd.20598. PMID 16400673
- [Background] Tublin ME, Bude RO, Platt JF. Review. The resistive index in renal Doppler sonography: where do we stand? AJR Am J Roentgenol. 2003 Apr;180(4):885-92. doi: 10.2214/ajr.180.4.1800885. No abstract available. PMID 12646425
- [Background] Vadas M. and Limaye v. 2005. The vascular endothelium: structure and function. In: Fitridge R. and Thompson M., editors. Mechanisms of Vascular Disease: A Textbook for Vascular Surgeons. Cambridge University Press: pp 1-10
- [Background] Waanders F, van Timmeren MM, Stegeman CA, Bakker SJ, van Goor H. Kidney injury molecule-1 in renal disease. J Pathol. 2010 Jan;220(1):7-16. doi: 10.1002/path.2642. PMID 19921716
- [Background] Waikar SS, Curhan GC, Wald R, McCarthy EP, Chertow GM. Declining mortality in patients with acute renal failure, 1988 to 2002. J Am Soc Nephrol. 2006 Apr;17(4):1143-50. doi: 10.1681/ASN.2005091017. Epub 2006 Feb 22. PMID 16495376
- [Background] Yalavarthy R, Edelstein CL. Therapeutic and predictive targets of AKI. Clin Nephrol. 2008 Dec;70(6):453-63. doi: 10.5414/cnp70453. PMID 19049701
- [Background] Yang L, Besschetnova TY, Brooks CR, Shah JV, Bonventre JV. Epithelial cell cycle arrest in G2/M mediates kidney fibrosis after injury. Nat Med. 2010 May;16(5):535-43, 1p following 143. doi: 10.1038/nm.2144. Epub 2010 May 2. PMID 20436483
- [Background] Liu Y. Renal fibrosis: new insights into the pathogenesis and therapeutics. Kidney Int. 2006 Jan;69(2):213-7. doi: 10.1038/sj.ki.5000054. PMID 16408108

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT05414669/Prot_SAP_ICF_000.pdf